CLINICAL TRIAL: NCT04974775
Title: Swecrit Biobank - Blood Samples From Critically Ill Patients and Healthy Controls
Acronym: SWECRIT
Status: Active, not recruiting | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Region Skane (Other); Lund University (Other)
Responsible Party: Principal Investigator, Hans Friberg, Professor, Consultant, Skane University Hospital
Other Study IDs: SWECRIT
Record Dates: First submitted 2021-06-18; First posted 2021-07-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-11

CONDITIONS: Critical Illness; Cardiac Arrest; Sepsis; Influenza; Covid19; Trauma
Keywords: Biobank; Critical Illness; Cardiac Arrest; Sepsis; Influenza; Covid-19; Trauma; Prognosis; Neurology
MeSH Terms: conditions — Critical Illness; Heart Arrest; Sepsis; Influenza, Human; COVID-19; Wounds and Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood, plasma, and serum are stored at -80°C in the biobank BD-47 at IDEON, Lund, Sweden.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Critically Ill: Critically ill patients and patients in need of post-operative intensive care.
  Interventions: Diagnostic Test: Blood collection
- Cardiac Arrest: Cardiac Arrest according to the ICD-10 I469 diagnosis.
  Interventions: Diagnostic Test: Blood collection; Diagnostic Test: Blood collection, serial sampling
- Sepsis: Sepsis according to the sepsis-3 criteria.
  Interventions: Diagnostic Test: Blood collection
- Covid-19: Critically ill patients with a positive Covid-19 test.
  Interventions: Diagnostic Test: Blood collection; Diagnostic Test: Blood collection, serial sampling
- Influenza: Critically ill patients with a positive influenza test.
  Interventions: Diagnostic Test: Blood collection
- Trauma: Critically ill patients after a severe traumatic event.
  Interventions: Diagnostic Test: Blood collection
- Healthy controls: Healthy at the time of blood sampling
  Interventions: Diagnostic Test: Blood collection

INTERVENTIONS:
Diagnostic Test: Blood collection — Sampling on admission to ICU (all patients)
Diagnostic Test: Blood collection, serial sampling — Additional sampling to admission samples in
  1. the Cardiac Arrest group after 12 and 48 hours
  2. the Covid-19 group on day 2 and 7 while in the ICU
  3. the Covid-19 group after 3 and 12 months.
  Groups: Cardiac Arrest; Covid-19

SUMMARY:
Blood samples are collected and stored in a biobank for later analysis of circulating substances in peripheral blood and genetic variations in patients with severe critical illness and risk of death. The aim is to analyze stored samples in order to identify substances that can help predict the outcome of critically ill patients, but also to optimize treatment and possibly prevent serious illness and death in the future.

DETAILED DESCRIPTION:
SWECRIT is a regional, multicenter study with prospective collection of blood samples and background information from critically ill patients, admitted to an Intensive Care Unit (ICU) in Region Skåne, Sweden. Patients were originally categorized into four study cohorts a) cardiac arrest, b) sepsis, c) influenza, and d) trauma. In April of 2020, a fifth study cohort, covid19, was added to the original ones. In addition, a control group of healthy controls has been enrolled.

Diagnoses, disease course, treatment results and survival are prospectively collected from all critically ill patients in the Patient Administrative System for Intensive Care Units (PASIVA). PASIVA is the portal by which collected laboratory and physiological data are entered into the Swedish Intensive Care Register (SIR). Further data are collected retrospectively from other health-related registers, such as the Swedish Population Register, the International Cardiac Arrest Registry (INTCAR), The Swedish CPR Registry, the Swedish Trauma Registry (SweTrau), and the Regional quality register Covid-IR (covid19 disease).

Specifically for the covid19-cohort, detailed face-to-face follow-up will be performed of all survivors at 3 & 12 months and a telephone interview after 3 years. Questionnaires (see below) will be sent to patients prior to the follow-up. Questions about well-being in general, quality-of-life, sleeping disorders, psychological and psychiatric problems will be addressed.

Collected blood samples in the ICU are processed by clinical chemistry at each participating hospital and frozen specimens of whole blood, serum, and plasma (200 ul aliquots) are sent to the biobank BD-47 in Region Skane for long-term storage (maximum 20 years).

The circulating substances and genetic markers, i.e. biomarkers that will be analyzed are: proteins (markers of inflammation, stress, infection, neurologic injury, myocardial injury and endothelial function) and other circulating substances in the blood (metabolomics), genes (DNA) from the entire genome, epigenetic changes (eg methylation status of DNA), gene fragments (eg secretory DNA), various forms of RNA such as micro-RNA & longcoding RNA.

Research questions for future analyzes of collected samples are specified but subject to change, depending on progress and development in the specific research field of each study cohort.

1. Identification and use of biomarkers for assessment of severity of disease and trajectory over time in the ICU will be the main area of research.
2. Assessment of neurological prognosis and outcomes will be a common denominator in several studies.
3. Descriptive statistics and regression analyses will be performed in order to identify independent variables (biomarkers) of importance for prognosis and outcomes.

Inquiries to access the sample collection for research purpose can be sent to the central contacts listed below.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients admitted to the ICU
* 18 years or older
* covid19-verified (covid19-cohort)

Exclusion Criteria:

* The patient or next of kin decline participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All critically ill patients admitted to the participating ICUs in Region Skane (2015-2018), and a healthy control group.
  Starting in May 2020, critically ill Covid-19 patients admitted to an ICU in the Skane Region are prospectively included.
Sampling Method: Probability Sample
Enrollment: 8500 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality (all) | 6 months
  Primary outcome when functional outcome cannot be assessed.

SECONDARY OUTCOMES:
Proportion of patients with good neurological outcome 1 (all) | 3-6 months
  Neurological outcome assessed using Cerebral Performance Category 1-5 (CPC 1-5), CPC 1 representing the best and CPC 5 the worst outcome. Good outcome is defined as CPC 1-2, poor outcome as CPC 3-5.
Proportion of patients with good neurological outcome 2 (all) | 3-6 months
  Modified Rankin Score 0-6 (mRS 0-6), mRS 0 representing the best and mRS 6 representing the worst outcome. Good outcome is defined as mRS 0-3, poor outcome as mRS 3-6.
Neurological outcome 3 (covid19) | 3-6 months
  Glasgow Outcome Scale Extended 1-8 (GOSE 1-8), GOSE 1 representing the worst outcome and GOSE 8 the best outcome.

OTHER OUTCOMES:
Severity of the Acute Respiratory Distress Syndrome (ARDS) (covid19) | On ICU admission
  Patients fulfilling the ARDS criteria are categorized into mild, moderate or severe, depending on the ratio of arterial oxygen partial pressure (mmHg) to fractional inspired oxygen (FiO2). Mild: < 300, Moderate: < 200, Severe: < 100.
Proportion of patients with pathological Pulmonary Function Testing (PFT) | 3 and 12 months
  A composite of Total Lung Capacity (TLC) & Diffusion capacity (DLCO) compared to a population norm. Less than 80 % of the (age-adjusted) population norm is considered pathological.
Subjective respiratory function (covid19) | 3, 12 and 36 months
  Saint George's Respiratory Questionnaire 0-100 (SGRQ 0-100), lower values representing better function and higher values representing worse function. 8.41 (SD 11.33) is considered a normative value (Spanish population).
Physical problems (covid19) | 3, 12 and 36 months
  Short form Health Survey, version 2, physical function 10 (SF-36 v.2 PF-10), 10 items, higher score for each item represents better function. Scores are transformed to T-scores based on norm-based values. A T-score of 50 indicates the norm mean for each item. At a group level scores <47 and individual scores <45 indicate low physical function.
Proportion of patients with significant Fatigue (covid19) | 3, 12 and 36 months
  Modified fatigue impact scale 0-84 (MFIS 0-84), higher values representing more fatigue and lower numbers representing less fatigue. A value >38 discriminates significant fatigue.
Hospital Anxiety and Depression Scale (covid19) | 3, 12 and 36 months
  Anxiety and depression. Two sub-scales with 7 items in each, higher values represent more anxiety and depression, >8 points in each sub-scale indicates significant symptoms of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Friberg, MD, PhD, Study Chair — Skane University Hospital
Locations (4):
- Sweden (4):
  - Helsingborg Hospital, Helsingborg
  - Kristianstad Central Hospital, Kristianstad
  - Skane University Hospital, Lund
  - Skane University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lengquist M, Lundberg OHM, Spangfors M, Annborn M, Levin H, Friberg H, Frigyesi A. Sepsis is underreported in Swedish intensive care units: A retrospective observational multicentre study. Acta Anaesthesiol Scand. 2020 Sep;64(8):1167-1176. doi: 10.1111/aas.13647. Epub 2020 Jun 18. PMID 32463121
- [Background] Lundberg OHM, Lengquist M, Spangfors M, Annborn M, Bergmann D, Schulte J, Levin H, Melander O, Frigyesi A, Friberg H. Circulating bioactive adrenomedullin as a marker of sepsis, septic shock and critical illness. Crit Care. 2020 Nov 4;24(1):636. doi: 10.1186/s13054-020-03351-1. PMID 33148300
- [Background] Thorgeirsdottir B, Levin H, Spangfors M, Annborn M, Cronberg T, Nielsen N, Lybeck A, Friberg H, Frigyesi A. Plasma proenkephalin A 119-159 and dipeptidyl peptidase 3 on admission after cardiac arrest help predict long-term neurological outcome. Resuscitation. 2021 Jun;163:108-115. doi: 10.1016/j.resuscitation.2021.04.021. Epub 2021 Apr 27. PMID 33930500
- [Background] Johnsson J, Bjornsson O, Andersson P, Jakobsson A, Cronberg T, Lilja G, Friberg H, Hassager C, Kjaergard J, Wise M, Nielsen N, Frigyesi A. Artificial neural networks improve early outcome prediction and risk classification in out-of-hospital cardiac arrest patients admitted to intensive care. Crit Care. 2020 Jul 30;24(1):474. doi: 10.1186/s13054-020-03103-1. PMID 32731878
- [Derived] Arctaedius I, Wasselius J, Lang M, Drake M, Johnsson M, Friberg H, Leithner C, Kenda M, Lybeck A, Moseby-Knappe M. The semi-quantitative cardiac arrest brain ischemia (CABI) score for magnetic resonance imaging predicts functional outcome after cardiac arrest. Crit Care. 2025 Aug 20;29(1):373. doi: 10.1186/s13054-025-05595-1. PMID 40836345
- [Derived] Didriksson I, Frigyesi A, Spangfors M, Leffler M, Reepalu A, Nilsson AC, Annborn M, Lybeck A, Friberg H, Lilja G. Long-term recovery in critically ill COVID-19 survivors: A prospective cohort study. Acta Anaesthesiol Scand. 2025 Jan;69(1):e14550. doi: 10.1111/aas.14550. PMID 39540322
- [Derived] Didriksson I, Lengquist M, Spangfors M, Leffler M, Sievert T, Lilja G, Frigyesi A, Friberg H, Schiopu A. Increasing plasma calprotectin (S100A8/A9) is associated with 12-month mortality and unfavourable functional outcome in critically ill COVID-19 patients. J Intensive Care. 2024 Jul 9;12(1):26. doi: 10.1186/s40560-024-00740-4. PMID 38982551
- [Derived] Arctaedius I, Levin H, Larsson M, Friberg H, Cronberg T, Nielsen N, Moseby-Knappe M, Lybeck A. 2021 European Resuscitation Council/European Society of Intensive Care Medicine Algorithm for Prognostication of Poor Neurological Outcome After Cardiac Arrest-Can Entry Criteria Be Broadened? Crit Care Med. 2024 Apr 1;52(4):531-541. doi: 10.1097/CCM.0000000000006113. Epub 2023 Dec 7. PMID 38059722